CLINICAL TRIAL: NCT04651179
Title: A Retrospective Observational Study of the Effectiveness of Gemcitabine -Docetaxel in Patients With Relapsed Osteosarcoma Who Have Been Treated With HD-IFO in First Line Treatment
Brief Title: Study of Effectiveness of GEMDOX in Relapsed Osteosarcoma
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Ospedale Infantile Regina Margherita Sant'Anna (Other)
Responsible Party: Principal Investigator, Prof. Franca Fagioli, Principal Investigator, Azienda Ospedaliera Ospedale Infantile Regina Margherita Sant'Anna
Other Study IDs: OSTEOREC/OSS
Record Dates: First submitted 2020-11-24; First posted 2020-12-03 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Osteosarcoma Recurrent; Osteosarcoma Metastatic
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observation — not applicable, observational study

SUMMARY:
A retrospective observational study of the effectiveness of gemcitabine - docetaxel in patients with relapsed osteosarcoma who have been treated with HD IFO in first line treatment

ELIGIBILITY:
Inclusion Criteria:

* Age at diagnosis of high grade osteosarcoma >= 4
* Received first line treatment with HD IFO
* Following HD IFO treatment, they have been diagnosed refractory disease and they satisfy at least one of the following criteria :

  1. Relapsed in the first 24 month following the initial diagnosis, regardless of location and resectability
  2. Lung relapsed disease with more than 2 nodules diagnosed over 24 months from the initial diagnosis
  3. Non resectable relapsed disease diagnosed over 24 months from the initial diagnosis Before or during GEMDOX treatment, eligible patients may have been subject to metastasectomy

Exclusion Criteria: none

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with relapsed osteosarcoma treated with gemcitabine- docetaxel after a first line with HD- IFO
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2020-04-24 (Actual); Primary Completion 2021-06-06 (Actual); Study Completion 2021-11-23 (Actual)

PRIMARY OUTCOMES:
Response to Gemcitabina - Docetaxel Treatment | 12 months
  assessed as overall survival (12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Franca Fagioli, MD, Principal Investigator — AOU Città della Salute e della Scienza di Torino - Presidio Infantile Regina Margherita
Locations (8):
- Italy (8):
  - Istituto Nazionale Tumori, Milan, Milano
  - Fondazione del Piemonte per l' Oncologia IRCCS Candiolo, Candiolo, Turin
  - Istituto Ortopedico Rizzoli, Bologna
  - AOUC Azienda Ospedaliero-Universitaria Careggi, Florence
  - IRCCS Istituto Nazionale dei Tumori, Milan
  - Azienda Ospedaliero Universitaria pisana, Pisa
  - IRCCS Istituti Fisioterapici Ospitalieri, Rome
  - AOU Città della Salute e della Scienza di Torino - Presidio Infantile Regina Margherita, Turin

IPD SHARING:
Plan to Share IPD: No